CLINICAL TRIAL: NCT04932980
Title: Study Comparing Early Extension of Aflibercept and Brolucizumab in Wet AMD (SPARROW)
Brief Title: Comparison of Rapid Aflibercept and Brolucizumab T&E in wAMD
Acronym: SPARROW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berner Augenklinik (Other)
Collaborators: medignition AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPARROW 2021-01236
Record Dates: First submitted 2021-06-06; First posted 2021-06-21 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: wAMD; Treat & Extend; Aflibercept; Brolucizumab; Loading-phase
MeSH Terms: interventions — aflibercept; brolucizumab

STUDY DESIGN:
Intervention Model Description: two-armed, randomized, double-blind
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aflibercept ® rapid treatment extension (T&E) (Active Comparator): Early treat and extend (T&E) with Aflibercept ®. First IVT followed by control after 3 weeks and 2nd IVT after 6 weeks (= shortest treatment interval). Treatment will be adjusted according to morphologic response by adaptation of treatment intervals in +/- two-week increments.
  Interventions: Drug: Aflibercept; Procedure: early treat and extend (T&E)
- Brolucizumab ® rapid treatment extension (T&E) (Active Comparator): Early treat and extend (T&E) with Brolucizumab ®. First IVT followed by control after 3 weeks and 2nd IVT after 6 weeks (= shortest treatment interval). Treatment will be adjusted according to morphologic response by adaptation of treatment intervals in +/- two-week increments.
  Interventions: Drug: Brolucizumab; Procedure: early treat and extend (T&E)

INTERVENTIONS:
Drug: Aflibercept — administration of anti-VEGF Aflibercept (Eylea)
  Arms: Aflibercept ® rapid treatment extension (T&E)
Drug: Brolucizumab — administration of anti-VEGF Brolucizumab (Beovu)
  Arms: Brolucizumab ® rapid treatment extension (T&E)
Procedure: early treat and extend (T&E) — extension of treatment intervals (T&E) from the beginning of treatment

SUMMARY:
The currently widely established and preferred protocol for the treatment of wet age-related macular degeneration includes a loading phase of three monthly injections without interim adaptation or treatment according to disease activity, thereafter following a T&E strategy with treatment adaptation in increments of 2-4 weeks according to disease activity. Based on pharmacological considerations regarding the vitreal half-life of the drugs, the aim of this prospective explorative study is to test whether an early extension of treatment intervals without a loading phase is an option without compromising functional outcomes. Based on a superiority of Afl compared to Ran with regard to achieving a dry retina after one year and based on studies, but in the absence of real-life experience with Bro, it seems of interest to test how far Afl and Bro are comparable in terms of their potential to extend the treatment intervals over 12 months, the time to dryness of the retina, and number of injections. Also, it is of high clinical relevance to demonstrate efficacy with longer initial treatment intervals compared to the current possibly over-treating loading-phase with three four-weekly injections.

ELIGIBILITY:
Inclusion Criteria:

* Active MNV secondary to nAMD, going along with clinically significant vision loss
* Patients aged 50 years or older of all sexes
* Presence of IRF and/or SRF and/or subretinal hyperreflective material affecting the central subfield of the study eye on OCT
* signed informed consent for this study prior to the screening visit
* If possible: availability of a smartphone and willingness to perform self-testing with the Alleye app (soft criteria)

Exclusion Criteria:

* Any other cause of macular oedema
* Structural damage to the macula precluding a visual potential
* Optical media opacities not allowing an accurate performance of the protocol examinations
* Any intraocular surgery within three months prior to inclusion and history of any vitreoretinal surgery
* Advanced diabetic retinopathy potentially requiring any treatment within six months following inclusion or history of vitreal haemorrhage
* Presence of vitreoretinal traction or tractive epiretinal membrane affecting the fovea
* History of IVT with anti-VEGF or corticosteroids at any time in the study eye
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc.
* Significantly worse functional prognosis in the other eye or only eye
* Women of childbearing potential not willing to use an effective method of contraception during treatment and until at least 3 months after the last treatment
* Pregnant or lactating women
* Any systemic auto-inflammatory and auto-immune disease requiring treatment
* Treatment with high-dose corticosteroids (Prednisone equivalent >5mg/day), immunosuppressive or immunomodulatory or anti-proliferative agents for any reason
* Inability or contraindications to undergo the investigated intervention

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of injections given until week 52 | 52 weeks
  number injections received by patient

SECONDARY OUTCOMES:
Injections until week 104 | 104 weeks
  number injections received by patient
Number of treatment failures | 52 weeks
  number with treatment demand of less than 6 weeks at any time point
Number of treatment failures | 104 weeks
  number with treatment demand of less than 6 weeks at any time point
Time until drying of retina | 52 weeks
  mean interval until absence of intra- and subretinal fluid
Time until drying of retina | 104 weeks
  mean interval until absence of intra- and subretinal fluid
portion of eyes without disease activity | 52 weeks
  % patients with absence of intra- and subretinal fluid
portion of eyes without disease activity | 104 weeks
  % patients with absence of intra- and subretinal fluid
eyes under treatment intervals of ≥12 weeks | 52 weeks
  portion of eyes with stable disease under treatment intervals of ≥12 weeks
eyes under treatment intervals of ≥12 weeks | 104 weeks
  portion of eyes with stable disease under treatment intervals of ≥12 weeks
Change in visual acuity | 52 weeks
  change of VA in logRAD from baseline to week 52
Change in visual acuity | 104 weeks
  change of VA in logRAD from baseline to week 104
Change in central subfield thickness (CST) | 52 weeks
  change from baseline to week 52
Change in central subfield thickness (CST) | 104 weeks
  change from baseline to week 104
Portion of eyes gaining and loosing ≥5, ≥10, and ≥15 letters | 52 weeks
  change from baseline to week 52
Portion of eyes gaining and loosing ≥5, ≥10, and ≥15 letters | 104 weeks
  change from baseline to week 104
Maximal treatment interval extension | 52 weeks
  mean treatment interval extension
Maximal treatment interval extension | 104 weeks
  mean treatment interval extension

CONTACTS AND LOCATIONS:
Overall Officials: Justus G. Garweg, Prof. Dr. med., Principal Investigator — Berner Augenklinik
Locations (1):
- Berner Augenklinik, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fauser S, Schwabecker V, Muether PS. Suppression of intraocular vascular endothelial growth factor during aflibercept treatment of age-related macular degeneration. Am J Ophthalmol. 2014 Sep;158(3):532-6. doi: 10.1016/j.ajo.2014.05.025. Epub 2014 May 28. PMID 24879948
- [Background] Garweg JG, Gerhardt C. Disease stability and extended dosing under anti-VEGF treatment of exudative age-related macular degeneration (AMD) - a meta-analysis. Graefes Arch Clin Exp Ophthalmol. 2021 Aug;259(8):2181-2192. doi: 10.1007/s00417-020-05048-1. Epub 2021 Feb 2. PMID 33528645